CLINICAL TRIAL: NCT00449228
Title: Evaluation of Preoperative Education and Mini-invasive Total Hip Replacement in Regard to the Attainment of Functional Independency and Reduction of Hospital Stay
Brief Title: Efficacy of Preoperative Education and Mini-invasive Surgery for Total Hip Replacement
Acronym: ANRACT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Cochin Hospital (Ambiguous)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P051040
Record Dates: First submitted 2007-03-18; First posted 2007-03-20 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2007-03

CONDITIONS: Osteoarthritis of the Hip
Keywords: Osteoarthritis,; hip replacement,; education,; randomized controlled trial,; mini-invasive surgery
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: -preoperative education and total hip replacement — -preoperative education and total hip replacement

SUMMARY:
We propose to evaluate a preoperative education of the patient and a new surgical technique (the mini-invasive THR) that could reduce the time to achieve functional independence.

The primary objective of the trial is to assess the time to reach functional independence after total hip replacement depending on the treatment groups: preoperative education versus no preoperative education and mini-invasive procedure versus standard procedure. The study hypothesis is that education and mini-invasive procedure will reduce the time to reach functional independence.

This is a prospective trial with a double randomization.

DETAILED DESCRIPTION:
We propose to evaluate a preoperative education of the patient and a new surgical technique (the mini-invasive THR) that could reduce the time to achieve functional independence. Preoperative education is compared to no education and the mini-invasive surgery is compared to the standard group.

The education is based on explaining to the patient what will the postoperative rehabilitation be like.

The mini-invasive THR is based on the minimisation of soft tissue trauma. It requires a specific instrumentation to allow dissection and implantation of the prosthesis. Only few studies have evaluated such a technique. However, these studies were retrospective or non-randomised and results are contradictory. Therefore, a randomised controlled clinical trial is necessary to evaluate the possible benefits and feasibility of this technique.

The primary outcome is the time to reach functional independence. Secondary outcomes evaluate the duration of hospital stay, the quality of implantation of the prosthesis, the postoperative morbidity, the functional benefits and the quality of life.

Methods: this monocentric randomised controlled clinical trial compares the preoperative education versus no preoperative education (first randomization) and the conventional THR to the mini-invasive THR (second randomization). One hundred and forty patients will be included in each group.

Expected results: preoperative education and the mini-invasive THR are prone to decrease time to functional independence, postoperative morbidity and duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the hip
* avascular necrosis of the hip
* patient between 40 and 90 years old (included)

Exclusion Criteria:

* history of previous hip operation (bone)
* patient >90 or < 40
* inflammatory arthritis
* important proximal femur or acetabular deformity
* complete functional independence not possible
* BMI > 30

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2007-04; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Time to reach functional independence at hospital discharge | during de study
  Time to reach functional independence at hospital discharge

SECONDARY OUTCOMES:
Perioperative criteria : | during the study
  Perioperative criteria :
estimated blood loss | during the study
  estimated blood loss
duration of operation | during the study
  duration of operation
implant position | during the study
  implant position
implant fixation | during th study
  implant fixation
perioperative technical errors | during the study
  perioperative technical errors
Postoperative during hospital stay: | during the study
  Postoperative during hospital stay:
number of patients and number of units transfused before hospital discharge | during the study
  number of patients and number of units transfused before hospital discharge
total estimated blood loss | during the study
  total estimated blood loss
postoperative pain | during the study
  postoperative pain
skin problems | during the study
  skin problems
duration of hospital stay | during the study
  duration of hospital stay
Postoperative (3, 6 and 12 months): | during the study
  Postoperative (3, 6 and 12 months):
Harris hip score, SF-36, evaluation of satisfaction and expectation | during the study
  Harris hip score, SF-36, evaluation of satisfaction and expectation
Abduction strength, balance and gate | during the study
  Abduction strength, balance and gate
Scar assessment | during the study
  Scar assessment
complications | during the study
  complications

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ANRACT, PU-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Cochin, Paris, France